CLINICAL TRIAL: NCT04560452
Title: A Multi-Centre, Prospective, Non-Interventional Study to Intensively Monitor the Safety of Olaparib in Clinical Practice Among Chinese Patients.
Brief Title: Drug Intensive Monitoring Study of Olaparib in Clinical Practice Among Chinese Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00011
Record Dates: First submitted 2020-09-07; First posted 2020-09-23 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Prostate Cancer
Keywords: OC and PC
MeSH Terms: conditions — Ovarian Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Prostate cancer: according to the doctor's decision, have prescribed and agreed to start taking at least one dose of Olaparib
- Ovarian cancer: At least take one tablet of olaparib before enrolment for OC cohort

SUMMARY:
This is a multi-centre, prospective, non-interventional study. The study will enrol about 860 Chinese cancer patients from around 56 sites. For OC cohort, the subjects who had received olaparib for at least one dose before study enrolment in real world practices will be enrolled ( n=800) . For PC cohort, according to the doctor's decision, patients who have prescribed and agreed to start taking at least one dose of Olaparib will be enrolled ( n=60). Patient's treating physician is in charge of prescribing (including dose-adjusting or interruption) or discontinuation of olaparib.

DETAILED DESCRIPTION:
The study will enrol about 1,000 Chinese cancer patients from around 56 sites. For OC cohort, the subjects who had received olaparib for at least one dose before study enrolment in real world practices will be enrolled ( n=800) . For PC cohort, according to the doctor's decision, patients who have prescribed and agreed to start taking at least one dose of Olaparib will be enrolled ( n=60). Patient's treating physician is in charge of prescribing (including dose-adjusting or interruption) or discontinuation of olaparib.

The recruited patients will be followed up according to standard clinical practice. They will be tracked up to 30 days after discontinuation of olaparib treatment, or 6 months for Cohort OC, 12 months for Cohort PC after enrolment.Every OC patient will be followed maximum of 6 months after enrolment as Olaparib AEs most occur in first 6m and PC patient will be followed maximum of 12 months to observe 1-year PFS. Any adverse events (AEs) that are ongoing at the patient's last visit in the study must be followed up by the investigator for as long as medically indicated, but without further recording in the electronic case report form (eCRF).

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
* Patients diagnosed as olaparib approved tumor types in China
* Eligible for olaparib treatment per the judgement of the treating physician in clinical practice
* For OC cohort: at least take one tablet of olaparib before enrolment
* For PC cohort: according to the doctor's decision, have prescribed and agreed to start taking at least one dose of Olaparib

Exclusion Criteria

• In other ongoing studies, which prohibit any participation in this non-interventional study judged by investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit about 1000Chinese cancer patients from around 56 sites in real world practice in approved tumor types.
Sampling Method: Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with AEs as well as number of AE events as assessed by CTCAE | from the time of signature of informed consent, throughout the treatment period and until the end of study follow-up, up to 6 months for Cohort OC, 12 months for Cohort PC after enrolment.
  The primary objective of this study is to describe the safety and tolerability of olaparib in Chinese patients by assessing the incidence, seriousness, causality, severity and action taken (interruption/dose reduction/discontinuation) of all AEs (including AESIs) among all enrolled patients (including OC and PC patients as a whole). The number and percentage of patients with AEs as well as number of AE events will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) preferred terms and Common Terminology Criteria for Adverse Events (CTCAE) grade.

SECONDARY OUTCOMES:
Number and percentage of patients with AEs as well as number of AE events as assessed by CTCAE | from the time of signature of informed consent, throughout the treatment period and until the end of study follow-up in special populations, up to 6 months for Cohort OC, 12 months for Cohort PC after enrolment.
  To describe the safety and tolerability of olaparib in special populations (including patients with hepatic impairment or renal impairment, elderly patients with age > 65 years old) in Chinese patients by assessing the incidence, seriousness, causality, severity and action taken (interruption/dose reduction/discontinuation) of all AEs (including AESIs) among enrolled special populations. The number and percentage of patients with AEs as well as number of AE events will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) preferred terms and Common Terminology Criteria for Adverse Events (CTCAE) grade for special populations.
Progression-free survival(PFS) for PC cohort | From the date of treatment initiation, until investigator-reported progression or death, up to 12 months.
  PFS will be measured as the date of treatment initiation, until investigator-reported progression or death due to any cause, whichever occurs first for PC cohort.
PFS rate at one year for PC cohort | From the date of treatment initiation, until investigator-reported progression or death, up to 12 months.
  PFS rate at one year is defined as the proportion of patients who are alive and progression free at 12 months after the start of treatment for PC cohort.
Time to treatment discontinuation(TTTD) for PC cohort | From the date of treatment initiation, until the earlier of the date of treatment discontinuation or death, up to 12 months.
  TTTD will be measured as the date of treatment initiation, until the earlier of the date of treatment discontinuation or death for PC cohort.
Number and percentage of patients with different treatment pattern for PC cohort | From the time of signature of informed consent, throughout the treatment period and until the end of study follow-up, up to 12 months.
  Number and percentage of patients with different treatment pattern,which will be classified by concomitant medications and procedures including surgery, radiation therapy, chemotherapy and hormone therapy (including castration therapy and anti-androgen therapy) for PC cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongqiu Lin, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (37):
- China (37):
  - Research Site, Anhui
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Fujian
  - Research Site, Guangdong
  - Research Site, Guangzhou
  - Research Site, Guangzho
  - Research Site, Guizhou
  - Research Site, Hangzhou
  - Research Site, He'nan
  - Research Site, Hebei
  - Research Site, Heilongjiang
  - Research Site, Henan
  - Research Site, Huizhou
  - Research Site, Jiangsu
  - Research Site, Jiangxi
  - Research Site, Jilin
  - Research Site, Jinghou
  - Research Site, Liaoning
  - Research Site, Luzhou
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Sichuan
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Yichang
  - Research Site, Yunan
  - Research Site, Zhejiang
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No